CLINICAL TRIAL: NCT04032561
Title: The Relationship Between the Elevation of Haemoglobin A1c Level, Sleep Quality and Sleep Duration in Clinically Diagnosed Pre-diabetic Patients in a Nationally Representative Sample
Brief Title: Relationship Between HbA1c Level, Sleep Quality and Sleep Duration
Status: Completed | Type: Observational
Sponsor: University of Hertfordshire (Other)
Responsible Party: Principal Investigator, Terun Desai, Lead Investigator, University of Hertfordshire
Other Study IDs: LMS/UG/NHS/02928
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus, Type 2; Pre Diabetes; Sleep Disorder
Keywords: HbA1c; Sleep Quality; Sleep Duration; PSQI
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will be conducted during the period of, January 2019 - August 2019 with pre-diabetic participants on a NHS England funded National Diabetes Prevention Program (NDPP) with a clinically diagnosed Haemoglobin A1c (HbA1c) referral reading of between 42mmol/mol - 47mmol/mol within the last 12 months. The term pre-diabetic can all be used to explain blood glucose levels that are higher than normal, but not high enough for participants to be diagnosed with Type 2 diabetes. Having high blood glucose levels can increase a participant's risk of developing Type 2 diabetes and other health complications, although this is not inevitable.

100 participants will take part in the study. Participants will be eligible if they are aged between 18 and 65 years and have an HbA1c referral reading of between 42-47mmol/mol within the last 12 months.

The participants will be given a written consent form to sign to take part in the study, after receiving both written and verbal information beforehand on the study protocol from the researcher. Health screening to determine eligibility for the NHS funded program will be undertaken directly by the intervention provider.

Study design and procedures:

The study will be delivered in a controlled format and will be designed to assess the relationship between the elevation of HbA1c level, sleep quality and sleep duration in clinically diagnosed pre-diabetic participants referred and registered to join the NHS NDPP. Participants will receive a pre-program information pack in conjunction with a sleep quality and sleep duration questionnaire at the end of their 1:1 initial appointments for the NHS NDPP.

Participants will be given prepaid envelopes to send their anonymised questionnaires back to the researcher once completed after their appointments. The researcher will ensure confidentiality by keeping all questionnaires in a securely combination coded locked cupboard that only the researcher has access to. Participants will be instructed to not write their names on the questionnaires but to only state their gender, age, and referral HbA1c reading received from the relevant health care professional.

ELIGIBILITY:
Inclusion Criteria:

* Participants were eligible if they were aged 18 years - 65 years
* Had an HbA1c referral reading of between 42-47mmol/mol within the last 12 months
* Registered on the NHSE NDPP

Exclusion Criteria:

* Participants with a severe debilitating disease which may have interfered with the study participation
* Under the age of 18 years or over the age of 65 years
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged 18 years - 65 years with pre-diabetes (diagnosed as HbA1c referral reading of between 42-47mmol/mol within the last 12 months)
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 1 month
  Sleep quality was measured from PSQI.
  Scoring system:
  Not during the past month = 0 Less than once a week = 1 Once or twice a week = 2 Three or more times a week = 3
Sleep Duration | 1 month
  Sleep duration was measured from PQSI.
  Scoring system:
  Not during the past month = 0 Less than once a week = 1 Once or twice a week = 2 Three or more times a week = 3

SECONDARY OUTCOMES:
HbA1c | Within 12 months
  Retrieved from NHS referral database

CONTACTS AND LOCATIONS:
Locations (1):
- NHS/HSC Site, London, United Kingdom